CLINICAL TRIAL: NCT01194687
Title: Reproducibility of a Fecal Occult Blood Test Device for Gut Microbiota Analyses
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910107; 10-C-N107
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09-14

CONDITIONS: Normal Physiology
Keywords: Estrogens; Fecal Microbiome; Fecal Occult Blood

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Bacteria and other micro-organisms in the intestines play important roles in immunity and other health conditions. As a result, these micro-organisms are likely to affect many health conditions, including several types of cancer. Because cancer and other diseases may affect the digestive system and the bacteria within it, fecal samples that are taken both before and after the onset of a disease may show important changes in the body and provide information about possible treatments. However, unlike repositories of blood and tissue samples, researchers do not have a repository of fecal specimens. Researchers are interested in determining whether standard collection procedures used for fecal occult blood testing can provide accurate information on micro-organisms in the intestine.

Objectives:

- To determine whether standard fecal occult blood testing procedures can provide accurate collections of fecal micro-organisms for research purposes.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* At the clinical center, participants will be provided with written and illustrated instructions for the collection procedures and a self-administered risk questionnaire. The questionnaire will assess the challenges of collecting fecal specimens and will collect data on major dietary restrictions (e.g., vegan, vegetarian, food allergies), medication use and major illnesses, knowledge of and past experience with fecal occult blood testing, colonoscopy and colon cancer, and the fecal collection devices.
* Participants will be provided with a collection bag for the sample, 16 sample collection tubes, and a box with frozen gel packs.
* On the morning of collection, participants will collect the fecal sample in the bag and use the collection tubes to obtain material from different parts of the stool.
* The tubes will be sealed and placed in the box with the gel packs, and the participant will hand deliver the entire box to the clinical center.
* Characteristics of the bacteria in the material will be measured by laboratories at the University of Maryland.
* Statistical comparisons will determine how well the procedures worked.

DETAILED DESCRIPTION:
Commensal bacteria and other microbial organisms (the microbiota), particularly in the intestines, are centrally related to nutrition, metabolism, immunity, inflammation, and endocrine balance. As an initial step toward possible establishment of a biobank of feces that could be used for prospective studies of the relationship of microbiota to cancer and other conditions, we propose a study to evaluate whether fecal microbiota, as well as microbial enzyme expression and function, are reproducibly represented in feces that has been collected with a device that is widely used for fecal occult blood testing (FOBT-CHEK oc). To do so, this study will recruit a convenience sample of 50 volunteers from DCEG and others at NIH. From a single stool, each participant will provide 16 aliquots of feces, half collected with FOBT-CHEK oc and the rest with a larger Sarstedt device. A urine sample and a brief self-administered questionnaire on antibiotics and other medications, serious chronic diseases, and major cancer risk factors will also be obtained. The aliquots will be used for microbiome pyrosequencing, beta-glucuronidase and beta-glucosidase expression and enzymatic activity. Variance within and between collection devices, as well as between individuals, will be quantified. This study will provide insight and quantitative estimates that will be required for formal studies of the relationship of the fecal microbiome to cancer. Under an amendment, to examine the ability of selected antibiotics to stabilize fecal microbial populations when they have been stored at 3 or 7 days prior to freezing, 10 of the same volunteer participants will be asked to provide aliquots of a second stool specimen. Differences between immediate and delayed freezing with or without the antibiotics will be tested by analysis of variance. Under an amendment, up to 100 participants will be enrolled to examine reproducibility of the microbiota with a used commercial colorectal cancer screening device and the stability of the microbiota within individuals over four years, participants will be asked to collect specimens during 2014, exactly as was done during 2010. Assays and anlyses will be analogous to those performed previously.

ELIGIBILITY:
* INCLUSION CRITERIA:

NIH employee, minimum age 18 years.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-04-27; Study Completion 2018-09-14

PRIMARY OUTCOMES:
Micriobiome Reproducibility | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Sinha, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Flores R, Shi J, Gail MH, Gajer P, Ravel J, Goedert JJ. Assessment of the human faecal microbiota: II. Reproducibility and associations of 16S rRNA pyrosequences. Eur J Clin Invest. 2012 Aug;42(8):855-63. doi: 10.1111/j.1365-2362.2012.02659.x. Epub 2012 Mar 3. PMID 22385292
- [Background] Flores R, Shi J, Gail MH, Ravel J, Goedert JJ. Assessment of the human faecal microbiota: I. Measurement and reproducibility of selected enzymatic activities. Eur J Clin Invest. 2012 Aug;42(8):848-54. doi: 10.1111/j.1365-2362.2012.02660.x. Epub 2012 Mar 13. PMID 22409163
- [Background] Flores R, Shi J, Fuhrman B, Xu X, Veenstra TD, Gail MH, Gajer P, Ravel J, Goedert JJ. Fecal microbial determinants of fecal and systemic estrogens and estrogen metabolites: a cross-sectional study. J Transl Med. 2012 Dec 21;10:253. doi: 10.1186/1479-5876-10-253. PMID 23259758